CLINICAL TRIAL: NCT06251349
Title: Comparative Analysis of Radiotherapeutic and Medical Procedures for the Prophylaxis of Heterotopic Ossifications in the Context of Total Hip Arthroplasty
Brief Title: Comparative Analysis of Radiotherapeutic and Medical Procedures for the Prophylaxis of Heterotopic Ossifications
Acronym: CONFIDENTIAL
Status: Completed | Type: Observational
Sponsor: University of Jena (Other)
Responsible Party: Principal Investigator, Matthias Mäurer, Principal Investigator, University of Jena
Other Study IDs: 2023-3175-Daten
Record Dates: First submitted 2024-01-22; First posted 2024-02-09 (Actual); Last update posted 2024-02-09 (Actual); Status verified 2024-02

CONDITIONS: Heterotopic Ossification; Hip Arthropathy; Myositis Ossificans Traumatica, Thigh
Keywords: Heterotopic Ossification; Total Hip Arthroplasty; Irradiation Hip; Diclofenac; Prevention of HO; NSAID; Brooker Classification
MeSH Terms: conditions — Ossification, Heterotopic | interventions — Radiation; Diclofenac

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Intervention group with prophylactic irradiation: Patients with total hip arthroplasty and irradiation (preoperative on the day before the operation (>24h preoperative)) Quantity: 128 Period: 01.01.2013 - 31.12.2023
  Interventions: Radiation: Radiation
- Control group with prophylactic NSAID-treatment: Patients with total hip arthroplasty and diclofenac treatment Quantity: 384 Period: 01.01.2013 - 31.12.2023
  Interventions: Drug: Diclofenac

INTERVENTIONS:
Radiation: Radiation — Single dose radiation with 7-8 Gy
  Groups: Intervention group with prophylactic irradiation
Drug: Diclofenac — postoperative treatment with diclofenac to prevent HO
  Other Names: NSAID-Treatment
  Groups: Control group with prophylactic NSAID-treatment

SUMMARY:
Aim of this study is to proof the efficacy of in Jena established prophylaxis of new bone formation aside the skeleton with irradiation and compare it with the common literature. Furthermore we want to compare irradiation treatment with the alternative prophylaxis with analgetics from the NSAID type.

DETAILED DESCRIPTION:
Aim of this retrospective analysis is to compare the incidence of heterotopic ossification one year after total hip arthroplasty with the at our location established concept of irradiation 24h preoperative and incidence in common literature. Furthermore the comparison between irradiated patients and patients treated with NSAIDs.

ELIGIBILITY:
Inclusion Criteria:

Patients with total hip arthroplasty performed at Eisenberg Patients with preoperative irradiation (24h pre-op) or postoperative diclofenac treatment Patients with x-ray images immediately (3-5 days postoperative) postoperative and at least 365 days postoperative

Exclusion Criteria:

Patients with missing follow up image

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All participants of the study are patients at the Universitätsklinikum Jena or the Waldkrankenhaus Eisenberg. Irradiation was performed in Jena. Total hip arthoplasty and following inpatient stay, inclusive NSAID therapy was performed in Eisenberg
Sampling Method: Non-Probability Sample
Enrollment: 512 (Actual)
Dates: Start 2013-01-01 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Presence of heterotopic ossification (HO) | at least 365 days postoperative
  X-ray controlled HO diagnostics with the Brooker classification

CONTACTS AND LOCATIONS:
Overall Officials: Matthias Mäurer, Dr., Study Director — Klinik für Strahlentherapie und Radioonkologie des Universitätsklinikums Jena
Locations (1):
- Department of Radiooncology, Jena, Jena, Germany

IPD SHARING:
Plan to Share IPD: No